CLINICAL TRIAL: NCT00473993
Title: Hepatitis C Bei Opioidabhängigen in Der Praxis, Eine Querschnittsuntersuchung
Brief Title: Hepatitis C Among Opioid Addicts in Opioid Maintenance Treatment in Zurich, Switzerland
Acronym: HepCOP
Status: Completed | Type: Observational
Sponsor: Seidenberg, Arztpraxis A., M.D. (Individual)
Collaborators: University of Zurich (Other)
Other Study IDs: HepCOP Zurich
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2007-05

CONDITIONS: Hepatitis C, Chronic; Substance Abuse Treatment Centers; Opioid-Related Disorders
Keywords: Hepatitis C; Opioid Maintenance Treatment; Methadone; Buprenorphine; Heroin; Interferon, pegylated
MeSH Terms: conditions — Hepatitis C, Chronic; Opioid-Related Disorders; Hepatitis C

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hepatitis C viral infection is common among opioid addicts in Zurich, Switzerland. The majority undergoes a maintenance treatment with methadone, heroin or buprenorphine. While stabilized by an opioid maintenance treatment (OMT)chronic hepatitis C can be treated with pegylated interferon plus ribavirin. As not sufficiently known, the results are comparable to the results of the treatment of nonaddicts.

Our crossectional study investigates how many patients undergoing OMT are adequately investigated concerning hepatitis C. If not, why are they not adequately investigated and treated? Representative data are collected in the local clinics and medical practices involved in OMT in the Kanton of Zurich. The patients files are revised and the involved doctors are asked through a structured interview.

DETAILED DESCRIPTION:
www.seidenberg.ch/hepcop.pdf

ELIGIBILITY:
Inclusion Criteria:

* Medical practices and clinics involved in opioid maintenance treatment in the Kanton of Zurich, Switzerland

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients in opioid maintenance treatment in the kanton of Zurich, Switzerland
Dates: Start 2007-07; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: André Seidenberg, Dr.med., Study Director — research fellow EHAM, University of Zurich

REFERENCES:
- See also: download of the protocol of the HepCOP-study — http://www.seidenberg.ch/media/hepcop.pdf